CLINICAL TRIAL: NCT02007473
Title: A Prospective Non-interventional Study to Evaluate the Safety of Methylene Blue Plasma
Status: Completed | Type: Observational
Sponsor: Maco Productions S.A.S. (Industry)
Collaborators: SynteractHCR (Industry)
Responsible Party: Sponsor
Other Study IDs: 1974/MCP
Record Dates: First submitted 2013-11-29; First posted 2013-12-10 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Adverse Effects in the Therapeutic Use of Plasma Substitutes
Keywords: Haemovigilance; Plasma; Pathogen reduction; Methylene Blue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients requiring transfusion with plasma: Recipients, who have received a transfusion with Methylene Blue plasma produced using the THERAFLEX MB-Plasma procedure from MacoPharma.

SUMMARY:
The objective of this non-interventional study is to gather data on adverse reactions occurring with Methylene Blue plasma administered in a routine clinical practice environment; to know more about their characteristics and behaviour and the possible factors that may influence their presentation and evolution.

DETAILED DESCRIPTION:
This is an open label, multi-centre, non-controlled, non-randomized, non-interventional study to evaluate the safety of Methylene Blue (MB) plasma. One centre per country will participate from United Kingdom, Belgium, Greece and Spain.

The haemovigilance Case Report Form (CRF) will be completed for all patients who receive a Methylene Blue plasma transfusion and experience an adverse reaction. The patients will be monitored for the occurrence of possible adverse reactions within 24 hours after start of the transfusion. If the patient experiences an adverse reaction, information about the adverse reaction will be documented. Serious adverse reactions will be collected within a 7-day period after the transfusion.

Each adverse reaction or serious adverse reaction will be followed up for 28 days after the occurrence of the reaction.

Each centre will provide the number of transfused Methylene Blue plasma units and the number of transfused Methylene Blue plasma patients every three months.

Information collected on the haemovigilance CRF will include:

* Details about the transfusion (transfused units, volume, other non-plasma blood components transfused)
* Details about the plasma (collected from whole blood, aphaeresis or both, filter using, type of reference used, illumination device model)
* Demographic data
* Transfusion history (including hospital department)
* History of previous transfusion reactions
* Details about the adverse reaction (date and time of reaction)
* Signs and symptoms and allocation to a diagnosis
* Classification of the adverse reaction (severity, imputability, non-serious or serious)
* Actions taken
* Outcome
* Time to recovery

ELIGIBILITY:
Inclusion Criteria:

* Patients, who have received a transfusion with Methylene Blue plasma produced using the THERAFLEX MB-Plasma procedure from MacoPharma and experience an adverse reaction.

Exclusion Criteria:

* Patients receiving transfusion with other plasma types during the same transfusion episode

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inpatients requiring plasma transfusion
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2013-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The incidence of transfusion reactions following administration of Methylene Blue Plasma based on the total number of transfusions administered | One year

SECONDARY OUTCOMES:
The incidence of specific transfusion reactions following administration of Methylene Blue plasma | One year
  The rate of the different type of adverse events registered along the time frame.

OTHER OUTCOMES:
Relationship between transfusion reaction types and indication, gender, age and severity | One year
  Analysis of factors that could be related to transfusion reactions

CONTACTS AND LOCATIONS:
Overall Officials: Hafiz Qureshi, MD, PhD, Principal Investigator — University Hospitals, Leicester; Mercedes Villamayor, MD, PhD, Principal Investigator — Complejo Hospitalario Universitario de Santiago; Lucien Noens, MD PhD, Principal Investigator — University Ghent; Aggeliki Megalou, MD PhD, Principal Investigator — G. H. A. Evaggelismos, Athens
Locations (4):
- Universitair Ziekenhuis, Ghent, Belgium
- G. H. A. Evaggelismos, Athens, Greece
- Complexo Hospitalario Universitario, Santiago de Compostela, La Coruña, Spain
- University Hospitals of Leicester NHS Trust, Leicester, United Kingdom